CLINICAL TRIAL: NCT07327801
Title: Impact of Ultrasound Guidance on the Performance of Spinal Anesthesia
Brief Title: The Impact of Ultrasound-Guided Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, askrihaythem, Associate Professor, Military Hospital of Tunis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 54/2024/clpp/militaryhosptunis
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Ultrasound Guidance; Spinal Anesthesia; Procedural Performance; Conventional Palpation Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional spinal anesthesia (Active Comparator): The operator began by palpating the posterior superior iliac spines to mentally determine the Tuffier's line, which roughly corresponds to the L4-L5 intervertebral space. The spinous processes were then palpated to precisely locate the targeted intervertebral space. The needle was subsequently inserted until cerebrospinal fluid return was obtained, and the anesthetic agent was administered slowly
  Interventions: Device: Conventional spinal anesthesia
- Ultrasound-guided spinal anesthesia (Active Comparator): The operator set up the sterile equipment, which included an ultrasound machine equipped with a low-frequency convex probe (2-5 MHz). The probe, previously disinfected, was covered with a sterile sheath containing sterile coupling gel.
  First, the transducer was positioned in a paramedian sagittal plane, placed 1-2 cm lateral to the spinous processes. The sacrum was identified as a flat, hyperechoic structure producing a marked acoustic shadow, serving as the starting landmark for identifying successive lumbar intervertebral spaces. By gradually sliding the transducer cephalad, the vertebral laminae appeared as hyperechoic lines alternating with their posterior acoustic shadows. The interlaminar spaces, located between two adjacent laminae, form true acoustic windows that allow visualization of the underlying neuraxial structures.
  The exploration continued until the intervertebral space deemed optimal for puncture was identified. The probe was then switched to a midline posit
  Interventions: Device: Ultrasound-guided spinal anesthesia

INTERVENTIONS:
Device: Conventional spinal anesthesia — The spinous processes were then palpated to precisely locate the targeted intervertebral space
  Arms: Conventional spinal anesthesia
Device: Ultrasound-guided spinal anesthesia — A combined sequence was used, beginning with a longitudinal paramedian scan, followed by a 90-degree rotation to obtain a transverse interspinous view. This allowed for the identification of the spinal canal, after which the puncture was performed using dynamic, out-of-plane guidance
  Arms: Ultrasound-guided spinal anesthesia

SUMMARY:
Neuraxial anesthesia is a commonly employed technique for subumbilical surgical procedures due to its effectiveness and safety profile. The advent of ultrasound technology has introduced the possibility of visualizing anatomical landmarks in real time, thereby facilitating more accurate and potentially safer subarachnoid punctures. This study aims to compare conventional spinal anesthesia, based on palpation, with ultrasound-guided spinal anesthesia, focusing on procedural ease and overall facilitation.

it's a prospective, single-center, randomized, single-blind study. We included patients aged 18 years or older, classified as ASA I or II, scheduled for elective surgery, and who provided written informed consent. Exclusion criteria included failed subarachnoid puncture, conversion to general anesthesia, or the occurrence of major intraoperative complications such as vasovagal episodes or cardiac rhythm disturbances. Participants were randomly assigned, based on a randomization table, into two groups: Group1 (traditional technique), in which spinal anesthesia was performed using the conventional palpation-based method for space localization; and Group2 (ultrasound-guided technique), in which spinal anesthesia was performed under real-time ultrasound guidance. The primary outcome was the total procedure time, measured in seconds from the end of skin antisepsis to the initiation of subarachnoid injection. Secondary outcomes included the number of puncture attempts, the number of needle redirections within the same interspace, the occurrence of procedural incidents, and postoperative complaints such as radicular pain, osseous contact pain, intraoperative paresthesias, and traumatic punctures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Classified as American Society of Anesthesiologists (ASA) physical status I or II.
* Scheduled for elective surgery under spinal anesthesia.
* Provided written informed consent.

Exclusion Criteria:

* Failed subarachnoid puncture.
* Conversion to general anesthesia.
* Occurrence of major intraoperative complications (e.g., vasovagal episodes, cardiac rhythm disturbances).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
procedure time | 60sec

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided